CLINICAL TRIAL: NCT03485378
Title: Assessment of Precision Irradiation in Early NSCLC and Interstitial Lung Disease (ASPIRE-ILD): A Phase II Trial
Brief Title: Assessment of Precision Irradiation in Early NSCLC and Interstitial Lung Disease
Acronym: ASPIRE-ILD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other); University of British Columbia (Other); Western University, Canada (Other)
Responsible Party: Principal Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASPIRE-ILD
Record Dates: First submitted 2018-03-07; First posted 2018-04-02 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer; Interstitial Lung Disease
Keywords: Stereotactic; Ablative; Radiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm: Stereotactic Ablative Radiotherapy (Experimental): Stereotactic ablative radiotherapy for early non-small cell lung cancer and interstitial lung disease
  Interventions: Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy — Stereotactic ablative radiotherapy for early non-small cell lung cancer and interstitial lung disease

SUMMARY:
This is a prospective phase II study of Stereotactic Ablative Radiotherapy (SABR) in patients with Non-Small Cell Lung Cancer (NSCLC) and co-existent Interstitial Lung Disease (ILD), to determine oncologic and toxicity outcomes. Patients will be divided into 3 separate cohorts based on the ILD-GAP index.

DETAILED DESCRIPTION:
For patients with ILD and concurrent early-stage lung cancer who are not candidates for surgery, data showing high rates of toxicity have led to a difficult clinical dilemma, since there are few alternate treatment options. The option of delivering no treatment whatsoever, which avoids any risk of treatment-related toxicity, is associated with a high risk of death due to the lung cancer itself.

Stereotactic ablative radiotherapy (SABR) is a newer radiotherapy approach which uses modern radiotherapy planning and targeting technologies to precisely deliver larger, ablative doses of radiotherapy. SABR has been associated with high rates of local control. A major advantage of SABR is that in general, the toxicity profile is very favorable, even in patients with substantial co-morbid conditions.

It is possible that currently-used doses and fractionations of SABR, when given with strict planning criteria to minimize the risk of lung toxicity, have only a modest risk of treatment-related toxicity and represent the best possible approach.

This study will examine SABR versus a historical control of untreated stage I non-small cell lung cancer with Overall survival (OS) as the endpoint. OS was selected as it objectively reflects the potential benefits of treatment (i.e. extended survival), the harms of treatment (grade 5 toxicity), and the natural history of the ILD disease process itself.

ELIGIBILITY:
Inclusion Criteria:

* Stage T1-2, N0, M0 (AJCC Staging, 8th Edition - i.e. tumor size ≤ 5 cm) prior to registration.
* Not a candidate for surgical resection, determined by any of the following:
* Consultation with a thoracic surgeon
* Discussion at Multidisciplinary Team (MDT) rounds with a surgeon present
* Patient refusal of surgery
* Pathologically (histologically or cytologically) proven diagnosis of non-small cell lung cancer (NSCLC) is not required, but strongly recommended.
* If the risk of biopsy is unacceptable, pathologic confirmation is not required providing there is growth over time on Computed Tomography (CT) imaging and/or Fluorodeoxyglucose (FDG) avidity that is strongly suggestive of a primary NSCLC.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3;
* Age ≥ 18;
* Life expectancy > 6 months
* Fibrotic interstitial lung disease of any subtype, as diagnosed by a respirologist/pulmonologist.

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (e.g., carcinomas in situ of the breast, oral cavity, or cervix are permissible); previous lung cancer, if the patient is disease-free for a minimum of 2 years is permitted.
* Prior thoracic radiotherapy
* Plans for the patient to receive other local therapy while on this study, except at disease progression;
* Plans for the patient to receive systemic therapy (including standard chemotherapy or biologic targeted agents), while on this study, except at disease progression. Patients are allowed to receive anti-fibrotic agents used in the treatment of IPF or non-IPF fibrotic ILD (e.g. nintedanib, pirfenidone), or steroids, if those are part of their current ILD treatment regimen. Other immunosuppressive drugs such as mycophenolate, azathioprine, cyclophosphamide, and rituximab must be stopped for 2 weeks prior and 2 weeks after treatment.
* Active pregnancy
* Concurrent administration of any drugs with known radiosensitive effects (e.g. Methotrexate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 4 years
  Time from enrollment to death from any cause

SECONDARY OUTCOMES:
Toxicity as measured by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 8 years
Progression-Free Survival | 8 years
Local Control as determined via radiographic evidence | 8 years
Cough Severity as reported by the participant via 10 cm analogue Cough Severity Scale | 8 years
  Cough severity will be reported by participants via a scale, where a score of 100 is no cough and a score of 0 is the worst cough ever.
Rates of Acute-Exacerbation of Idiopathic Pulmonary Fibrosis (IPF) | 8 years
Rates of Acute-Exacerbation of ILD | 8 years
Quality of Life measured by the Functional Assessment of Cancer Therapy - Lung questionnaire | 8 years
  The Functional Assessment of Cancer Therapy - Lung (FACT-L ) is a standardized questionnaire used to measure quality of life. The questionnaire consists of 5 scales measuring 37 items in total. Categories of the 5 scales are: physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns related to symptoms, cognitive function, and regret of smoking. The score for each item in the scale ranges from 0 to 4, where 0 is not at all and 4 is very much. The scores from each scale are added up, and can be combined to provide a total score.
Changes in ILD Severity measured by High Resolution Computed Tomography (HRCT) | 8 years
Changes in Pulmonary Function Tests | 8 years
Exploratory Quantitative Analysis of High Resolution Computed Tomography (HRCT) Features | 8 years
Analysis of Outcomes for Patients Eligible for Study Who Decline Radiotherapy | 8 years
Quality of Life measured by the EuroQOL Group EQ-5D-5L questionnaire | 8 years
  The EQ-5D-5L is a standardized questionnaire used to measure quality of life and health. The first section includes 5 categories: mobility, self-care, usual activities (e.g. work, family), pain/discomfort, and anxiety/depression. Each category contains 5 statements ranging from no problems to extreme problems, where no problems is assigned a code of 1 and extreme problems is assigned a code of 5. Participants are asked to select the statement that best describes their health that day. No score is generated, rather a 5 digit code is generated based on the response provided, which can then be combined into a data set and interpreted in a variety of ways. The second section includes a 20 cm analogue scale from 0 to 100, where 100 is the best health ever imagined and 0 is the worst health imagined. The participant will mark a score on the scale representing the state of their health on that day.

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, Study Chair — London Health Sciences Centre, Lawson Health Research Institute; Alexander Louie, MD, Study Chair — London Health Sciences Centre, Lawson Health Research Institute; Chris Ryerson, MD, Study Chair — University of British Columbia
Locations (6):
- Canada (5):
  - Alberta Health Services, Cross Cancer Institude, Edmonton, Alberta
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - UHN Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM Université de Montréal, Montreal, Quebec
- Edinburgh Cancer Centre, Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palma DA, Bahig H, Hope A, Harrow S, Debenham BJ, Louie AV, Vu TTTT, Filion E, Bezjak A, Campeau MP, Duimering A, Giuliani ME, Laba JM, Lang P, Lok BH, Qu XM, Raman S, Rodrigues GB, Goodman CD, Gaede S, Morisset J, Warner A, Dhaliwal I, Ryerson CJ. Stereotactic Radiation Therapy in Early Non-Small Cell Lung Cancer and Interstitial Lung Disease: A Nonrandomized Clinical Trial. JAMA Oncol. 2024 May 1;10(5):575-582. doi: 10.1001/jamaoncol.2023.7269. PMID 38451491
- [Derived] Palma DA, Chen H, Bahig H, Gaede S, Harrow S, Laba JM, Qu XM, Rodrigues GB, Yaremko BP, Yu E, Louie AV, Dhaliwal I, Ryerson CJ. Assessment of precision irradiation in early non-small cell lung cancer and interstitial lung disease (ASPIRE-ILD): study protocol for a phase II trial. BMC Cancer. 2019 Dec 11;19(1):1206. doi: 10.1186/s12885-019-6392-8. PMID 31829203